CLINICAL TRIAL: NCT06911996
Title: Immersive Bedside Teaching for Hospitalized Pediatric Patient - A Prospective, Mixed-method, Cohort Study
Brief Title: The WOW Project (WOW): Wonders Of The World Through Virtual Reality for Hospitalized Children
Acronym: WOW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 80079
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Virtual Reality
Keywords: Immersive Learning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual Reality Group (Experimental): Participants will all receive the VR intervention and will be instructed to wear an Oculus Quest 3 headset (Meta, Inc., Menlo Park, CA) and participate in virtual field trips from Engage (David Whelan). Brink Traveler (Akin Bilgic) and Wander (John Entwistle) that are specifically designed to reignite the joy and awe of learning.
  Interventions: Behavioral: Virtual Reality

INTERVENTIONS:
Behavioral: Virtual Reality — After obtaining written consent, participants will be asked to complete a brief demographic survey and pre-intervention surveys (content knowledge, and wellbeing surveys). They will then be equipped with a VR headset, Quest 3 (Meta, Inc., Menlo Park, CA) displaying the educational field trip. After the VR field trip, participants will participate in a complementary hands-on science experiment. At the conclusion of the experiment, patients will be asked to complete the post intervention surveys (i.e awe, content knowledge, and wellbeing surveys).
  Additionally, for the first 20 participants, 15 participants will be randomly selected and asked to participate in a 5 open-ended question qualitative interview regarding engagement of the lesson. Audio will be recorded via zoom.

SUMMARY:
Hospitalized pediatric patients are unable to leave the hospital to engage in traditional learning environments. Patients often feel depressed, disconnected from learning, and socially withdrawn. The Stanford Chariot Program proposes a partnership with the Palo Alto Unified Hospital School at Stanford Children's Health to reignite patients' emotional well-being through learning. The WOW Project aims to use virtual reality (VR) to travel with hospitalized children to the Wonders of the World (WOW). Combining this immersive learning modality with complementary hands-on activities at the bedside, the investigators will transport them from their hospital room into a nurturing virtual environment to stimulate their emotional, mental, and social growth while they are physically healing. The investigators will evaluate their overall joy and awe of learning by using standardized emotional scales.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 5 and 17.
* English speaking.
* Anticipated in-patient stay for more than 1 day.

Exclusion Criteria:

* Legal guardian not present to obtain consent
* Child with a significant neurological condition, or major developmental disability
* Child with active infection of the face or hand
* A history of severe motion sickness
* A history of seizures caused by flashing light
* Major surgery within the last 12 hours

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Assess the impact of VR-based field trips on the feeling of awe of the pediatric inpatient population | immediately after intervention
  The primary outcome will be AWE measured by the AWE-SF Survey - The Awe Experience Short Form Scale. The survey contains 12 items about awe experience. Each item was rated on a 7-point scale (1 = Strongly Disagree, 7 = Strongly Agree).

SECONDARY OUTCOMES:
Change in the number of correct answers of the content knowledge | Day 1 baseline, Day 1 immediately after intervention
  Change in number of correct answers of the content knowledge using Bloom's Taxonomy questioning. Participants will respond to 5 questions, two questions about comprehension, one question about application, one question about analysis and one question about evaluation. Scores range from 0 to 5, with higher scores indicating the higher number of correct answer.
Change in a patients' well-being as measured through the World Health Organization-Five Well-Being Index (WHO-5) | Day 1 baseline, Day 1 immediately after intervention
  The WHO (Five) Well-Being Index is a participant-reported outcome measure that assesses current mental well being. Questionnaire contains 5 questions . Scores range from 0 to 5, with higher scores indicating the corresponding feeling exists all the time.
Thematic analysis of the qualitative surveys including how the lesson engagement correlates to the increase in joyful learning. | immediately after intervention
  Analysis of data collected via qualitative surveys, using saturation sampling and documented coding techniques, will result in thematic descriptions how the lesson engagement correlates to the increase in joyful learning.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No